CLINICAL TRIAL: NCT05877261
Title: 5 Year Follow-Up of Migration of a Cementless Total Knee Replacement
Brief Title: Cementless Triathlon 5YR Follow-Up
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Schulich School of Medicine and Dentistry (Unknown)
Responsible Party: Principal Investigator, Brent Lanting, Orthopaedic Surgeon, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 12925
Record Dates: First submitted 2023-04-04; First posted 2023-05-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Knee Arthroplasty, Total; Knee Osteoarthritis; Radiostereometric Analysis
Keywords: Osteoarthritis; Cementless Fixation; Gut Microbiome; Weight-Bearing Computed Tomography
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Microbial DNA will be extracted from stool samples for 16s rRNA sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prior Cementless Knee Replacement Cohort: Patients who received a cementless knee replacement in 2017-2018 and participated in a prior study measuring the first year of implant migration.
  Interventions: Device: Cementless Total Knee Replacement

INTERVENTIONS:
Device: Cementless Total Knee Replacement — Artificial knee implant inserted by cementless fixation.

SUMMARY:
All artificial joint implants need to be solidly held (fixed) within the bone. Cementless fixation has become a popular method to achieve fixation for total knee replacements where the bone grows directly onto the implanted device instead of using bone cement. The primary purpose of this study is to assess long-term implant survivorship and clinical outcomes of a previous study cohort that received a cementless knee replacement. As this study cohort approaches 5 years post-operation, the investigators will re-examine the stability of participant implants using specialized x-rays, called "radiostereometric analysis". The study will use weight-bearing computed tomography (CT) to measure bone density and texture features and correlate that with implant stability. The investigators will collect stool samples to assess participant gut microbiomes for biomarkers of poor bone quality that could correlate to implant stability. All 33 participants from the original study cohort will be invited to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Were in the originally investigated cohort
* Had successful imaging at 1-year post-operation
* Minimum of 5 years post-operation

Exclusion Criteria:

* Pregnancy
* Unable to follow-up

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a cementless total knee replacement in 2017-2018 and participated in a previous study measuring the first year of implant migration.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Implant Migration (tibial component) | 5 year follow-up
  Implant movement will be measured with model-based Radiostereometric Analysis (RSA) by registering the location of the tibial component during supine exams. Potential tibial component migration between 1 and 5 years post-operation will be measured in millimeters with the use of tibial bone markers.

SECONDARY OUTCOMES:
Implant Migration (femoral component) | 5 year follow-up
  Implant movement will be measured with model-based Radiostereometric Analysis (RSA) by registering the location of the femoral component during supine exams. Potential femoral component migration between 1 and 5 years post-operation will be measured in millimeters with the use of femoral bone markers.
Inducible Displacement (RSA-based) | 5 year follow-up
  Model-based Radiostereometric Analysis (RSA) will be used to register the location of the tibial and femoral components during supine and standing exams. Change in implant position will be measured in millimeters as maximum total point motion (MTPM) between the standing and supine RSA exams.
Inducible Displacement (CT-based) | 5 year follow-up
  Weight-bearing computed tomography (CT) will be used to register the location of the tibial and femoral components during seated and standing exams. Change in implant position will be measured in millimeters as maximum total point motion (MTPM) between the seated and standing CT exams.
Bone Density | 5 year follow-up
  Weight-bearing computed tomography (CT) scans will be used to measure bone density as Hounsfield units in standardized volumes of interest below the pegs and keel of the tibial component.
Texture Features | 5 year follow-up
  Weight-bearing computed tomography (CT) texture analysis will be performed in standardized volumes of interest below the pegs and keel of the tibial component.
Microbial Diversity | 5 year follow-up
  Participants will provide a stool sample. Microbial DNA will be extracted from the stool samples for 16s rRNA sequencing. Taxonomy will be assigned and functional annotation will be determined.

OTHER OUTCOMES:
12-Item Short Form Survey (SF-12) | 5 year follow-up
  Patient reported outcome measure observing physical and mental health status of patient. There are 12 questions asking about health (excellent to poor), activity limitations (yes, limited a lot to no, not limited at all), problems with daily activities from physical or emotional health (yes or no), pain interfering with normal work (not at all to extremely), recent positive or negative feelings (all of the time to none of the time), and interference of physical or emotional problems with social activities (all of the time to none of the time). A higher score indicates better physical and mental health function.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 5 year follow-up
  Patient reported outcome measure observing physical symptoms following recent knee replacement surgery. Contains 24 questions asking about the amount of pain, stiffness, and activity difficulty (none to extreme). A higher score indicates greater pain, stiffness, and activity difficulty.
Knee Society Score (KSS) | 5 year follow-up
  Patient reported outcome measure. Contains 5 sections measuring patient symptoms (none to severe), satisfaction (very satisfied to very dissatisfied), expectation (too high to too low), functional activities, and discretionary knee activities. Functional activities are split into walking and standing (with or without aids and the duration), standard activities (no bother to cannot do), and advanced activities (no bother to cannot do). Discretionary knee activities measure difficulty with the three most important activities for the patient (no bother to cannot do). Higher scores indicate greater patient outcomes.
UCLA Activity Score | 5 year follow-up
  Patient reported outcome measure observing activity level of patient. Contains a 10-level scale with 1 representing a patient who is inactive and dependent on others, to 10 representing a patient who regularly participates in impact sports. A higher score indicates a greater activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, MD MSc FRCSC, Principal Investigator — Schulich School of Medicine and Dentistry
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddiqi A, Levine BR, Springer BD. Highlights of the 2021 American Joint Replacement Registry Annual Report. Arthroplast Today. 2022 Jan 29;13:205-207. doi: 10.1016/j.artd.2022.01.020. eCollection 2022 Feb. No abstract available. PMID 35128013
- [Background] Cherian JJ, Banerjee S, Kapadia BH, Jauregui JJ, Harwin SF, Mont MA. Cementless total knee arthroplasty: a review. J Knee Surg. 2014 Jun;27(3):193-7. doi: 10.1055/s-0034-1374811. Epub 2014 Apr 24. PMID 24764231
- [Background] Nam D, Lawrie CM, Salih R, Nahhas CR, Barrack RL, Nunley RM. Cemented Versus Cementless Total Knee Arthroplasty of the Same Modern Design: A Prospective, Randomized Trial. J Bone Joint Surg Am. 2019 Jul 3;101(13):1185-1192. doi: 10.2106/JBJS.18.01162. PMID 31274720
- [Background] Nam D, Bhowmik-Stoker M, Mahoney OM, Dunbar MJ, Barrack RL. Mid-Term Performance of the First Mass-Produced Three-Dimensional Printed Cementless Tibia in the United States as Reported in the American Joint Replacement Registry. J Arthroplasty. 2023 Jan;38(1):85-89. doi: 10.1016/j.arth.2022.07.020. Epub 2022 Aug 5. PMID 35934187
- [Background] Valstar ER, Nelissen RG, Reiber JH, Rozing PM. The use of Roentgen stereophotogrammetry to study micromotion of orthopaedic implants. ISPRS journal of photogrammetry and remote sensing 2002;56(5):376-89.
- [Background] Canadian Joint Replacement Registry. Hip and Knee Replacements in Canada: CJRR Annual Statistics Summary, 2018-2019.; 2019.
- [Background] Pijls BG, Plevier JWM, Nelissen RGHH. RSA migration of total knee replacements. Acta Orthop. 2018 Jun;89(3):320-328. doi: 10.1080/17453674.2018.1443635. Epub 2018 Mar 6. PMID 29508661
- [Background] Williams HA, Broberg JS, Howard JL, Lanting BA, Teeter MG. Effect of gap balancing and measured resection techniques on implant migration and contact kinematics of a cementless total knee arthroplasty. Knee. 2021 Aug;31:86-96. doi: 10.1016/j.knee.2021.05.011. Epub 2021 Jun 10. PMID 34119998
- [Background] Broden C, Sandberg O, Olivecrona H, Emery R, Skoldenberg O. Precision of CT-based micromotion analysis is comparable to radiostereometry for early migration measurements in cemented acetabular cups. Acta Orthop. 2021 Aug;92(4):419-423. doi: 10.1080/17453674.2021.1906082. Epub 2021 Apr 6. PMID 33821746
- [Background] Das M, Cronin O, Keohane DM, Cormac EM, Nugent H, Nugent M, Molloy C, O'Toole PW, Shanahan F, Molloy MG, Jeffery IB. Gut microbiota alterations associated with reduced bone mineral density in older adults. Rheumatology (Oxford). 2019 Dec 1;58(12):2295-2304. doi: 10.1093/rheumatology/kez302. PMID 31378815
- [Background] Ma R, Wu M, Li Y, Wang J, Yang P, Chen Y, Wang W, Song J, Wang K. The use of bone turnover markers for monitoring the treatment of osteoporosis in postmenopausal females undergoing total knee arthroplasty: a prospective randomized study. J Orthop Surg Res. 2021 Mar 17;16(1):195. doi: 10.1186/s13018-021-02343-3. PMID 33731168
- [Background] Al KF, Bisanz JE, Gloor GB, Reid G, Burton JP. Evaluation of sampling and storage procedures on preserving the community structure of stool microbiota: A simple at-home toilet-paper collection method. J Microbiol Methods. 2018 Jan;144:117-121. doi: 10.1016/j.mimet.2017.11.014. Epub 2017 Nov 16. PMID 29155236